CLINICAL TRIAL: NCT05744297
Title: NLRP3 Inflammasome Activation Among Patients During Acute Gout Flares
Acronym: ActiNG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ActiNG
Record Dates: First submitted 2023-02-02; First posted 2023-02-27 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-02

CONDITIONS: Gout Arthritis
MeSH Terms: conditions — Arthritis, Gouty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood and synovial fluid obtained from remainder of samples collected during standard of care required during acute goute flare.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gout is a chronic joint disease associated with deposition of monosodium urate crystals, as a consequence of hyperuricemia. Gout is an intermittent flaring condition and acute gout flares are driven by NLRP3 inflammasome and IL1-beta production.

However pathogenesis of acute gout flares remains poorly known in vivo in human.

The aim of this study is to evaluate NLRP3 inflammasome activation in vivo in patients cells during acute gout flares.

DETAILED DESCRIPTION:
Blood and synovial fluid will be obtained from remainder of patients' samples during an acute gout flares. White blood cells will be isolated and NLRP3 inflammasome activation will be assessed. Then, NLRP3 inflammasome inhibitors will be tested on cells with NLRP3 inflammasome activity.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for acute gout flare confirmed by joint fluid analysis or Nijmegen score > 8
* Aged > 18

Exclusion Criteria:

* Gout treatment already started
* Inflammatory Arthritis other than Gout Arthritis
* Pregnant or breast feeding women
* Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will be proposed to patients meeting study's criteria
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
NLRP3 inflammasome activation in white blood cells. | Patient admission at hospital
  White blood cells will be isolated from blood sample and NLRP3 inflammasome activation will be assessed by flow cytometry.

SECONDARY OUTCOMES:
NLRP3 inflammasome activation in synovial cells. | Patient admission at hospital
  Nucleated cells will be isolated from synovial fluid sample and NLRP3 inflammasome activation will be assessed by flow cytometry.
Effects of NLRP3 inflammasome inhibitors on proportion of NLRP3 inflammasome activation in white blood cells/synovial cells | up to 7 days after analysis of NLRP3 activity
  NLRP3 inflammasome inhibitors will be tested on cells with NLRP3 inflammasome activity in blood or synovial fluid.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Saint Joseph Saint Luc, Lyon, France

IPD SHARING:
Plan to Share IPD: No